CLINICAL TRIAL: NCT05255315
Title: Apport du Lambeau Libre antébrachial Dans la Reconstruction Post-exentération
Brief Title: Impact of Forearm Free Flap in Orbital Exenteration Reconstruction
Acronym: REXOR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Other Study IDs: IC-2020-19
Record Dates: First submitted 2022-02-14; First posted 2022-02-24 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Cancer
Keywords: Forearm free flap; Orbital exenteration; Temporalis muscle flap; Quality of life
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Comparative analysis comparing the morbidity of the antebrachial free flap to that of the temporal flap flap during exenteration as well as the rate of fitting patients with epithesis. — A retrospective analysis will be performed by comparing the computerized data of patients reconstructed with a free antebrachial flap to that of patients reconstructed with a temporal muscle flap.
  Another analysis, this time prospective, will be carried out by comparing the answers to the reconstruction specific questionnaires as well as the POSAS scores of patients reconstructed with either a free antebrachial flap or a temporalis muscle flap.

SUMMARY:
Orbital exenteration is the en bloc removal of the entire orbital contents. This mutilating surgical technique is reserved for the management of certain malignant orbito-palpebral tumors or those that secondarily invade the orbit.

Several types of exenteration have been described, more or less extended to the adjacent structures, with sometimes mixed ENT-neurosurgical approaches for lesions invading the endocranium and causing large losses of substance.

Different surgical reconstruction techniques have been developed over the years, from spontaneous epithelialization to free osteo-muscular flap and temporal muscle transpositions.

Reconstruction after exenteration is essential to limit the sequelae and to allow the patient who has undergone this trauma to regain social interactions, a quality of life and an optimal self-image.

The use of an antebrachial free flap would allow a faster healing and thus an earlier rehabilitation.

The main objective of the study was to compare the morbidity of the antebrachial free flap with that of the temporal flap during exenteration and the rate of fitting of patients with epitheses.

DETAILED DESCRIPTION:
Reconstruction after exenteration is essential to limit the after-effects and to allow the patient who has suffered this trauma to regain social interaction, quality of life and self-image.

The principal investigator hypothesize that reconstruction with a free antebrachial flap can improve the quality of life of an exentered patient while maintaining a low risk of intra- and post-operative morbidity.

The aim of such a study will therefore be to provide assistance to both surgeons and patients, as to the choice of the technique of orbital reconstruction, by highlighting objectively and subjective evidence of the benefits of one technique over the other.

The patients included in this study will have to answer two questionnaires, submitted by post or directly at the follow-up consultation. This study therefore falls within the framework of studies of minimal or moderate risk studies. They will be informed by telephone interview beforehand or directly in the consultation about the method of writing the questionnaires and their content.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were exentered and then reconstructed by free antebrachial flap or temporal muscle flap muscle flap at the Institut Curie Paris, between January 2005 and December 2020.

Exclusion Criteria:

* Legally protected patients
* Patients unable to give consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who were exentered and then reconstructed by free antebrachial flap or temporal muscle flap muscle flap at the Institut Curie Paris, between January 2005 and December 2020.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-11-10 (Estimated); Study Completion 2022-11-10 (Estimated)

PRIMARY OUTCOMES:
Temporal muscle flap patient questionnaire. | Baseline
  A questionnaire of quality of life and side effects related to surgery for patients having a temporal muscle flap reconstruction (13 questions with binary or numerical answers)
Antebrachial flap patient questionnaire | Baseline
  A questionnaire of quality of life and side effects related to surgery for patients having antebrachial flap reconstruction (17 questions with binary or numerical answers)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine DUBRAY-VAUTRIN, MD, Principal Investigator — Institut Curie
Locations (1):
- Institut Curie, Paris, France